CLINICAL TRIAL: NCT00878566
Title: Alberta Clinical Trial in Optimizing Hypertension: The RxAction Study
Brief Title: Alberta Clinical Trial in Optimizing Hypertension
Acronym: RxAction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ross T. Tsuyuki, Dr., University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005300
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
Keywords: hypertension; pharmacists; rural health; prescribing
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care
- Enhanced pharmacist care (Experimental)
  Interventions: Other: Enhanced pharmacist care

INTERVENTIONS:
Other: Enhanced pharmacist care — The primary intervention will be enhanced pharmacist care. Pharmacists will assess patients with regards to cardiovascular risk reduction including reviewing BP control, treatment goals and determining lifestyle modifications for the patient to undertake to help manage their BP. The pharmacist will also review the patient's current hypertensive therapy regimen and decide on the options for improvement of BP control (lifestyle modification, increase dose, additional BP medications), and implementation of these strategies.
  Other Names: Treatment group
  Arms: Enhanced pharmacist care
Other: Usual Care — Patients randomized to usual care will receive a wallet card for BP readings, pamphlet on BP and usual pharmacist and physician care. Patients will be seen at 12 weeks for interim BP measurement only. Both groups of patients will be seen at 24 weeks for BP measurement.
  Other Names: Control
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate the effect of enhanced pharmacist care (patient identification, assessment, education, prescribing/titration of antihypertensive medications and close follow-up) on systolic blood pressure (BP) reduction in patients with poorly controlled hypertension in the community setting.

DETAILED DESCRIPTION:
The study is a randomized, controlled trial of enhanced pharmacist care, with the unit of randomization as the patient. Participants will be randomized to enhanced pharmacist care (patient identification, assessment, education, close follow-up and prescribing/titration of antihypertensive medications or usual care. Participants will be patients in Alberta with undiagnosed or uncontrolled BP as defined by the Canadian Hypertension Education Program. The primary intervention will be enhanced pharmacist care. Pharmacists will assess patients with regards to cardiovascular risk reduction including reviewing BP control, treatment goals and determining lifestyle modifications for the patient to undertake to help manage their BP. The primary outcome will be a comparison of difference in change in systolic BP between enhanced care and usual care at 24 weeks follow-up. Secondary outcomes include the number of patients at their BP target at 24 weeks, number of new antihypertensive medication starts, number of antihypertensive dosage changes, number of antihypertensive medication changes and number of new prescriptions for ASA and cholesterol medications.

ELIGIBILITY:
Inclusion Criteria:

1. Overall average (after 2 visits) systolic ≥180 OR diastolic ≥110 mmHg in undiagnosed patients without macrovascular target organ damage, diabetes or chronic kidney disease
2. Overall average (after 2 visits) systolic ≥140 OR diastolic ≥90 for patients with undiagnosed hypertension with macrovascular target organ damage (coronary artery disease, cerebrovascular disease, DM)
3. In patients with diagnosed hypertension, systolic ≥140 (≥ 130 with DM or CKD) OR diastolic ≥90, (≥ 80 with DM or CKD)
4. Overall average (after 5 visits, for those without macrovascular target organ damage, DM, or CKD and without an existing hypertension diagnosis) systolic ≥140 OR diastolic ≥90 mmHg
5. Overall average (after 7 days of twice-daily home blood pressure monitoring , for those without macrovascular target organ damage, DM, or CKD and without an existing hypertension diagnosis) systolic ≥135 OR diastolic ≥85

Exclusion Criteria:

* Patients with hypertensive urgency or emergency:

  * Urgency: SBP ≥ 180 mm Hg or DBP ≥ 120 mm Hg with no acute signs of end-organ damage
* Unwilling to participate/sign consent form
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2009-11; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Comparison of difference in change in systolic BP between enhanced care and usual care | 24 weeks

SECONDARY OUTCOMES:
number of patients at their BP target | 24 weeks
number of new antihypertensive medication starts | 24 weeks
number of antihypertensive dosage changes | 24 weeks
EQ-5D | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ross T. Tsuyuki, PharmD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Tsuyuki RT, Houle SK, Charrois TL, Kolber MR, Rosenthal MM, Lewanczuk R, Campbell NR, Cooney D, McAlister FA; RxACTION Investigators*. Randomized Trial of the Effect of Pharmacist Prescribing on Improving Blood Pressure in the Community: The Alberta Clinical Trial in Optimizing Hypertension (RxACTION). Circulation. 2015 Jul 14;132(2):93-100. doi: 10.1161/CIRCULATIONAHA.115.015464. Epub 2015 Jun 10. PMID 26063762
- [Derived] Charrois TL, McAlister FA, Cooney D, Lewanczuk R, Kolber MR, Campbell NR, Rosenthal M, Houle SK, Tsuyuki RT. Improving hypertension management through pharmacist prescribing; the rural Alberta clinical trial in optimizing hypertension (Rural RxACTION): trial design and methods. Implement Sci. 2011 Aug 11;6:94. doi: 10.1186/1748-5908-6-94. PMID 21834970